CLINICAL TRIAL: NCT05603624
Title: Effect of Sterile Versus Clean Gloves Intrapartum and Postpartum Infections at Term
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Futility due to sample size needed to prove superiority and lack of difference in outcomes between intervention and control group.
Sponsor: Eastern Virginia Medical School (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 21-09-FB-0206
Record Dates: First submitted 2022-10-28; First posted 2022-11-02 (Actual); Last update posted 2023-08-25 (Actual); Status verified 2023-08

CONDITIONS: Chorioamnionitis; Intrauterine Infection; Postpartum Endometritis; Puerperal Infection
Keywords: Sterile glove; Clean glove; Glove type; Intraamniotic infection; Cervical examination; Sterile vaginal examination; Intrapartum infection; Postpartum infection
MeSH Terms: conditions — Chorioamnionitis; Puerperal Infection

STUDY DESIGN:
Intervention Model Description: Eligible and consented participants were randomized to receive all cervical examinations with sterile powder-free polyvinyl chloride exam gloves (current routine practice, control group) or clean powder-free nitrile exam gloves (nonsterile, experimental group). Neither the clinical providers performing the exam nor the participants were blinded to the glove type used, however, the researchers did not know which glove type was used while completing the retrospective data collection and analysis. All other obstetrical care provided to the participants was per ACOG guidelines and the only changes made to their care was the type of glove used for this study.
Who Masked: Investigator, Outcomes Assessor
Masking Description: The two types of gloves used were labeled as "Glove 1" and "Glove 2" for data collection and analysis. The providers performing examinations and the patients knew the type of glove being used at the time of the study but data collection was deidentified and retrospective analysis was blinded to the investigating team until the study concluded.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Sterile glove (Active Comparator): Sterile glove is usually the standard of care
  Interventions: Procedure: Cervical examination to assess labor
- Clean glove (Experimental): Clean glove is usually not used or in the event of an emergency or lack of access to sterile gloves in the United States.
  Interventions: Procedure: Cervical examination to assess labor

INTERVENTIONS:
Procedure: Cervical examination to assess labor — Patients were randomized to receive cervical examinations to assess progression in labor with either sterile or clean gloves.

SUMMARY:
This prospective randomized controlled study examines whether the type of glove used (sterile vs clean) for cervical examination to assess progression in labor impacts the rates of intrapartum and/or postpartum infection in patients during labor or induction of labor at term.

DETAILED DESCRIPTION:
Introduction The vaginal microbiota consists of a wide array of possible bacteria including species Ureaplasma, Listeria, Lactobacillus, Atopbium, Megasphaera, Leptotrichia, Peptostreptococcus, Prevotella, Diphtheria, Escherichia, Klebsiella, Enterobacter, Proteus, Pseudomonas, Gardnerella, Staphylococcus, and Streptococcus.1,2 However, the uterus is thought to be much less diverse in flora and possibly sterile, especially in the setting of pregnancy.3 Thickening of the cervical mucus functions as a buffer to prevent the polymicrobial vaginal bacteria from ascending into the uterus in pregnancy. Intraamniotic or intrauterine infections (IAI), also known as chorioamnionitis, are thought to occur most frequently from an ascending infection from the lower genital tract into the uterine cavity.4 IAI usually warrants immediate delivery and impacts 5 - 12% of term pregnancies, with the most commonly identified pathogenic species being Ureaplasma.5-7 IAI carries significant neonatal morbidity including increased risk for neonatal pneumonia, bronchopulmonary dysplasia, poor neonatal growth, dermatitis, necrotizing enterocolitis, retinopathy of prematurity, cerebral palsy, meningitis, sepsis, and death.4,7 When performing cervical examinations during labor, providers in the United States commonly use a sterile glove to examine dilation and effacement of the cervix and station of the fetal head, although there are no data currently to support that this practice reduces rates of infection. Even though the uterus could be sterile in normal pregnancies, the provider performing the cervical examination must traverse the milieu of diverse vaginal bacteria in order to reach the cervix to perform the exam, introducing vaginal microbiota into the uterus. Despite this, it is unclear if the number of cervical examinations impacts risk of infection, especially before rupture of membranes (ROM).8,9 Common risk factors for IAI acknowledged by the American College of Obstetrics and Gynecology (ACOG) include excessive number of cervical examinations (especially after rupture of membranes), cervical insufficiency, internal fetal heart rate or uterine contraction monitors, intracervical balloon catheters for induction of labor, urogenital pathogens (sexually transmitted infections (STI), group B streptococcus (GBS) colonization, bacterial vaginosis), nulliparity, alcohol and tobacco use in pregnancy, and meconium-stained amniotic fluid.4 Nevertheless, some of these factors are also associated with longer duration of labor, rupture of membranes, and more cervical examinations, so they may not be independently associated with IAI.8,10 The theory behind IAI, assuming there are no other sources of maternal infection present elsewhere that could be introduced into the uterus or passed through the placenta, is that an infection ascends from the vagina into the intrauterine or intraamniotic space to cause the infection. We hypothesize that the type of glove used for examination should not impact rates of intrapartum or postpartum infection since the glove, whether originally sterile or not, would have to pass through the unsterile vagina to reach the cervix to perform the cervical examination. This prospective randomized controlled study examines whether the type of glove used (sterile vs clean) impacts the rates of IAI in patients receiving cervical examinations during labor or induction of labor at term.

Methods Patients meeting the inclusion and exclusion criteria below provided written informed consent to participate in the study after admission to labor and delivery at the single institution tertiary care referral center for this study. Any cervical examinations performed prior to the patient being consented to participate in the study were not included, such as if performed in the office or in the triage area, prior to admission.

This study followed the format of a randomized prospective cohort study where eligible and consented participants were randomized to receive all cervical examinations with sterile powder-free polyvinyl chloride exam gloves (current routine practice, control group) or clean powder-free nitrile exam gloves (nonsterile, experimental group). Neither the clinical providers performing the exam nor the participants were blinded to the glove type used, however, the researchers did not know which glove type was used while completing the retrospective data collection and analysis. All other obstetrical care provided to the participants was per ACOG guidelines and the only changes made to their care was the type of glove used for this study.

Interested participants were eligible to participate if their pregnancy was at term (37w0d to 41w6d gestational age), if their amniotic membranes were intact on admission, if they were presenting in spontaneous labor or were to undergo induction of labor, and if they were attempting for a vaginal delivery initially, even if the final delivery method was by cesarean section. Participants were excluded if they were preterm (before 37w0d gestational age), postdates (after 41w6d gestational age), with ruptured membranes or premature rupture of membranes on admission, in preterm labor, with the diagnosis of chorioamnionitis or any intrauterine infection, with extrauterine infection that would compromise the diagnosis of intrauterine infection (e.g., COVID, upper respiratory infections, urinary tract infections, cellulitis, appendicitis, etc.), experiencing an immunocompromised state (e.g., human immunodeficiency virus, congenital syndromes, transplant recipient, or immunosuppressant use), with uncertainty of their gestational age or no prenatal care, with an intrauterine fetal demise, or requesting a termination of the pregnancy. Twin or multigestational pregnancies were not excluded, however, only singleton pregnancies consented to participate in the study.

The primary outcome of the study was the proportion of participants in each glove group who experienced intraamniotic or intrauterine infection or chorioamnionitis or intrapartum infection, these terms are used interchangeably for the purposes of this study. The diagnostic criteria for intraamniotic/intrauterine infection followed the ACOG committee opinion 7124 on the topic, listed below for reference:

Patients must have fever >39.0*C (102.2F) ONE TIME without need to recheck temperature in the presence of no other identifiable source of fever OR

Fever of 38.0 - 38.9*C (100.4 - 102.02F) on two or more measurements that are at least 30 minutes apart without another clear source PLUS one or more of the following:

* Baseline fetal heart rate >160 beats/min for ≥10 minutes, excluding accelerations, decelerations, and periods of marked variability.
* Maternal white cell (WBC) count >15,000/mm^3 in the absence of corticosteroids and ideally showing a left shift (bandemia).
* Purulent-appearing fluid coming from the cervical os visualized by speculum examination.

The study's secondary outcomes and other data recorded included:

Rates of endometritis, maternal age, gravida, parity, induction of labor (IOL) method (foley balloon, cook catheter or cervical ripening balloon, Cytotec (misoprostol), Pitocin (oxytocin), Dilapan, Cervidil), artificial or spontaneous rupture of membrane time (AROM and SROM respectively), time of first cervical exam, number of documented cervical exams, delivery time, delivery method (cesarean section vs vaginal delivery), operative delivery (forceps or vacuum), postpartum hemorrhage (qualitative blood loss > 1000 mL), GBS colonization, gestational diabetes mellitus (GDM), Type 1 or Type 2 diabetes mellitus (T1DM or T2DM, respectively), genitourinary infections (urinary tract infections (UTI), pyelonephritis, gonorrhea (Gc), chlamydia (Ch), trichomonas (Tr), or pelvic inflammatory disease), tobacco/alcohol/drug use in pregnancy, meconium stained fluid, intrauterine pressure catheter (IUPC) use, fetal scalp electrode (FSE) use, epidural use, length of IOL (first cervical exam to delivery time), starting dilation, initial white blood cell (WBC) level on presentation, initial maternal temperature, highest maternal temperature, initial maternal heart rate (HR), highest maternal HR, and fetal tachycardia, if present and noted in the maternal chart.

Participants were considered GBS colonized if they had a positive rectovaginal culture by polymerase chain reaction (PCR) during routine prenatal care. All patients with a GBS positive status received antibiotics per ACOG recommendations. GBS negative or participants that did not have a GBS rectovaginal culture were not considered GBS colonized in this study to help distinguish those participants receiving antibiotics in labor.

Statistical analysis and sample size:

Given that the estimated rates of IAI in term pregnancy is estimated to be between 5-12%, weekly analysis was performed to ensure that interim rates of infection did not exceed 20%, which is double the median expected rate at term and would warrant discontinuation of the study. Data was collected in a deidentified manner from chart review and input into a REDCap database for analysis. The study was approved by the Eastern Virginia Medical School Institutional Review Board under IRB 21-09-FB-0206.

Descriptive statistics were used to describe the demographic and baseline characteristics of each cohort. Independent group comparisons were used to assure that the randomization resulted in equal groups at baseline. Continuous variables were compared with a two-sample independent group t test for normally distributed data or by Wilcoxon-Mann-Whitney test for non-normally distributed continuous variables. For categorical variables, the two groups were compared by Chi square test or Fisher exact test based on expected cell size.

ELIGIBILITY:
Inclusion Criteria:

* Between 18 and 50 years old
* Term pregnancy (37w0d to 41w6d gestational age)
* Amniotic membranes were intact on admission
* Patient presenting in spontaneous labor or were to undergo induction of labor
* Patient attempting for a vaginal delivery initially, even if the final delivery method was by cesarean section

Exclusion Criteria:

* Preterm pregnancy (before 37w0d gestational age)
* Postdate pregnancy (after 41w6d gestational age)
* Ruptured membranes or premature rupture of membranes on admission
* Patient being evaluated for preterm labor
* Patient has diagnosis of chorioamnionitis or any intrauterine infection
* Patient has an extrauterine infection that would compromise the diagnosis of intrauterine infection (e.g., COVID, upper respiratory infections, urinary tract infections, cellulitis, appendicitis, etc.)
* Patient experiencing an immunocompromised state (e.g., human immunodeficiency virus, congenital syndromes, transplant recipient, or immunosuppressant use)
* Patient with uncertainty of their gestational age and/or no prenatal care
* Patient with an intrauterine fetal demise
* Patient requesting a termination of the pregnancy

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 163 (Actual)
Dates: Start 2021-09-02 (Actual); Primary Completion 2022-09-01 (Actual); Study Completion 2022-09-01 (Actual)

PRIMARY OUTCOMES:
Chorioamnionitis or intraamniotic or intrauterine infection | Through study completion, usually withing 72 hours after admission to labor and delivery
  As defined by ACOG committee opinion 712

SECONDARY OUTCOMES:
Postpartum endometritis | Through study completion, usually withing 72 hours after admission to labor and delivery
  As defined by ACOG committee opinion 712

CONTACTS AND LOCATIONS:
Overall Officials: Stacy Slat, MD, Principal Investigator — Eastern Virginia Medical School
Locations (1):
- Eastern Virginia Medical School, Norfolk, Virginia, United States

IPD SHARING:
Plan to Share IPD: Yes
If contacted, can share deidentified participant data.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: After analysis and upon request; for undetermined amount of time.
Access Criteria: If contacted, can share deidentified participant data.

REFERENCES:
- [Result] Lamont RF, Sobel JD, Akins RA, Hassan SS, Chaiworapongsa T, Kusanovic JP, Romero R. The vaginal microbiome: new information about genital tract flora using molecular based techniques. BJOG. 2011 Apr;118(5):533-49. doi: 10.1111/j.1471-0528.2010.02840.x. Epub 2011 Jan 20. PMID 21251190
- [Result] Larsen B, Monif GR. Understanding the bacterial flora of the female genital tract. Clin Infect Dis. 2001 Feb 15;32(4):e69-77. doi: 10.1086/318710. Epub 2001 Feb 9. PMID 11181139
- [Result] Perez-Munoz ME, Arrieta MC, Ramer-Tait AE, Walter J. A critical assessment of the "sterile womb" and "in utero colonization" hypotheses: implications for research on the pioneer infant microbiome. Microbiome. 2017 Apr 28;5(1):48. doi: 10.1186/s40168-017-0268-4. PMID 28454555
- [Result] Committee Opinion No. 712: Intrapartum Management of Intraamniotic Infection. Obstet Gynecol. 2017 Aug;130(2):e95-e101. doi: 10.1097/AOG.0000000000002236. PMID 28742677
- [Result] Rouse DJ, Landon M, Leveno KJ, Leindecker S, Varner MW, Caritis SN, O'Sullivan MJ, Wapner RJ, Meis PJ, Miodovnik M, Sorokin Y, Moawad AH, Mabie W, Conway D, Gabbe SG, Spong CY; National Institute of Child Health And Human Development, Maternal-Fetal Medicine Units Network. The Maternal-Fetal Medicine Units cesarean registry: chorioamnionitis at term and its duration-relationship to outcomes. Am J Obstet Gynecol. 2004 Jul;191(1):211-6. doi: 10.1016/j.ajog.2004.03.003. PMID 15295368
- [Result] Sweeney EL, Dando SJ, Kallapur SG, Knox CL. The Human Ureaplasma Species as Causative Agents of Chorioamnionitis. Clin Microbiol Rev. 2016 Dec 14;30(1):349-379. doi: 10.1128/CMR.00091-16. Print 2017 Jan. PMID 27974410
- [Result] Cahill AG, Duffy CR, Odibo AO, Roehl KA, Zhao Q, Macones GA. Number of cervical examinations and risk of intrapartum maternal fever. Obstet Gynecol. 2012 Jun;119(6):1096-101. doi: 10.1097/AOG.0b013e318256ce3f. PMID 22617572
- [Result] Gluck O, Mizrachi Y, Ganer Herman H, Bar J, Kovo M, Weiner E. The correlation between the number of vaginal examinations during active labor and febrile morbidity, a retrospective cohort study. BMC Pregnancy Childbirth. 2020 Apr 25;20(1):246. doi: 10.1186/s12884-020-02925-9. PMID 32334543
- [Derived] Morshedi B, Strohm S, James H, Springer C, Gould L, Thurman A, Slat S. Effect of sterile vs clean gloves for cervical checks in labor on maternal infection at term: a randomized trial. Am J Obstet Gynecol MFM. 2023 Jun;5(6):100931. doi: 10.1016/j.ajogmf.2023.100931. Epub 2023 Mar 24. PMID 36965695